CLINICAL TRIAL: NCT04662398
Title: Using of Testes' Shocker in Treating Sexual Disease and Dysfunction
Brief Title: Using of Testes' Shocker in Improving Sexual Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hashim Talib Hashim, Medical Student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HT98
Record Dates: First submitted 2020-11-28; First posted 2020-12-10 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Sexual Dysfunction; Sexual Abstinence; Sexual Desire Disorder; Erectile Dysfunction; Erectile Dysfunction Following Radical Prostatectomy; Erectile Dysfunction Following Cryotherapy; Erectile Dysfunction With Diabetes Mellitus; Erectile Dysfunction Following Radiation Therapy; Erectile Dysfunction Following Urethral Surgery; Erectile Dysfunction With Type 2 Diabetes Mellitus
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexual Abstinence; Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Case control
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case (Testes shocker device) (Active Comparator): The shocker will be used in delivering the current gradually on the testes and penis to improve the blood flow and stimulates the sexual activity among males.
  Interventions: Device: JT Device
- Control (non testes shocker device) (Sham Comparator): These groups will not given the shocks, shame device will be used instead and then compare the two results.
  Interventions: Device: JT Device

INTERVENTIONS:
Device: JT Device — Shocker giving electrical shocks on testes
  Other Names: Testes shocker

SUMMARY:
Using of testes' shocker in treating the sexual dysfunction.

DETAILED DESCRIPTION:
Using of electrical shocks in treating sexual dysfunction in males, rectile dysfunction and inability to perform sexually good.

ELIGIBILITY:
Inclusion Criteria:

* All patients with sexual dysfunction or erectile dysfunction

Exclusion Criteria:

* Patients with trauma or other causes that make them inactive sexually

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Sexual desire | less than one month
  improving the desire of sex by using the electric shocks directly on the testes and penis. This will be assessed by a questionnaire (validated and reliable) to assess their ability to have sex more actively or not.
Erectile dysfunction | less than one month
  solving the problem of erectile dysfunction and this will be assessed by examination and experience to see if there is an effect for the electric shocks on erectile improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Al Imam, MD, Principal Investigator — University of Mosul
Locations (1):
- Hashim Talib Talib Hashim, Nasiriyah, Thi Qar, Iraq

IPD SHARING:
Plan to Share IPD: No